CLINICAL TRIAL: NCT00684359
Title: Platelet Reactivity After Cessation of Clopid in the Setting of Coronary Stent Implantation I: PRACTICE I
Acronym: PRACTICE I
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Ron Waksman, MD, MedStar Research Institute/Cardiovascular Research Institute
Other Study IDs: PRACTICE I
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Disease
Keywords: Patients having PCI with a drug eluting stent
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Single center randomized parallel group study to determine if:

1. there is a temporary increase in platelet reactivity after abrupt discontinuation of clopidogrel due to a potential rebound phenomenon.
2. the effect of sudden discontinuation of clopidogrel 6 months post coronary angioplasty with adjunct drug eluting stent implantation compared to 12 month continuation of clopidogrel on platelet reactivity. And the association with MACE up to 12 months post coronary angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, > 18 years of age,
* Patients who are scheduled for an elective PCI with a drug eluting stent
* Patients willing to return for all required follow up visits.
* Patients live/work within a 60 mile radius of the Washington Hospital Center.

Exclusion Criteria:

* Patient has experienced an acute myocardial infarction within the preceding 48 hours of the subsequent angioplasty.
* Unprotected left main coronary disease with >50% stenosis;
* Patients with renal failure requiring dialysis;
* Patients with a documented ejection fraction < 30 percent at the time of subsequent PCI;
* Patient with a life expectancy less than 12 months or malignancy.
* Known allergies to aspirin or clopidogrel bisulfate (PlavixR) and that cannot be medically managed;
* Planned surgery or other indication for requiring the cessation of clopidogrel within 12 months of PCI;
* Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study.
* Patients with known history of bleeding diathesis;
* Prothrombin time >1.5 times control; coumadin therapy
* Platelet count <100 000/mm3;
* Hematocrit <25%;
* Creatinine >4.0 mg/dL;
* Thienopyridine use within 5 days of enrollment
* Glycoprotein (GP) IIb/IIIa use within 8 hours of enrollment or any indication were the operator will require GP IIb/IIIa inhibitor use during the hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, male or female, > 18 years of age; who are scheduled for an elective PCI with a drug eluting stent; willing to return for all required follow up visit and live/work within a 60 mile radius of the Washington Hospital Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-06; Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine if there is a temporary increase in platelet reactivity after abrupt discontinuation of clopidogrel due to a potential rebound phenomenon | Up to 12 months

SECONDARY OUTCOMES:
To determine what the effect of sudden discontinuation of clopidogrel 6 months post coronary angioplasty with adjunct drug eluting stent implantation compared to 12 month continuation of clopidogrel on platelet reactivity. | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ron Waksman, MD, Washington Hospital Center, Washington D.C., District of Columbia, United States